CLINICAL TRIAL: NCT04756856
Title: Impact of a Muscle-targeted Nutritional Therapy in the Recovery of Post-discharge COVID19 Patients Suffering From Sarcopenia
Brief Title: Muscle-targeted Nutritional Therapy for the Recovery From COVID-19
Acronym: RE-COVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant change in the profile of recruitable patients
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Emanuele Cereda, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210006520
Record Dates: First submitted 2021-02-15; First posted 2021-02-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Muscle-target oral nutritional supplementation (Experimental): Two servings (40 grams each) of powder (Fortifit; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, and 800 IU vitamin D
  Interventions: Other: Muscle-target oral nutritional supplementation

INTERVENTIONS:
Other: Muscle-target oral nutritional supplementation — Patients will receive daily for 12 weeks two servings (40 grams each) of powder (Fortifit; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, and 800 IU vitamin D. Patients will be also followed for 12 weeks after the suspension of supplementation.

SUMMARY:
To assess the impact of a muscle-targeted nutritional therapy consisting of nutritional counseling and high-quality whey protein-based oral nutritional supplements enriched with leucine and vitamin D, on the recovery of post-COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* Sarcopenia (revised European Working Group on Sarcopenia in Older People criteria)
* Recent discharge from hospital for COVID-19
* Informed consent

Exclusion Criteria:

* Any malignant disease during the last five years
* Known kidney failure (previous glomerular filtration rate <30 ml/min);
* Known liver failure (Child B or C)
* Psychiatric disease
* Endocrine disorders associated with disorders of calcium metabolism (excluding osteoporosis)
* Indications related to the study product:

More than 10 µg (400 IU) of daily Vitamin D intake from medical sources. More than 500 mg of daily calcium intake from medical sources. Adherence to a high energy or high protein diet up or use of protein containing or amino acid containing nutritional supplements up to three months before starting the study.

* Known allergy to milk, milk products or other components of the proposed interventions
* Indication to or ongoing artificial nutrition support
* Inclusion in other nutrition intervention trials
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Physical performance - chair-stand | 12 weeks
  Change in chair-stand test

SECONDARY OUTCOMES:
Physical performance - chair-stand | 24 weeks
  Change in chair-stand test at the end of study
Total body muscle mass | 24 weeks
  Change in total body muscle mass during the study
Appendicular muscle mass | 24 weeks
  Change in appendicular muscle mass during the study
Functional status - muscle strength | 24 weeks
  Change in handgrip strength during the study
Fatigue | 24 weeks
  Change in fatigue as assessed by the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) during the study
Energy intake | 24 weeks
  Change in energy intake during the study
Self-perceived quality of life | 24 weeks
  Change in quality of life during the study as assessed by the five-level EuroQol five-dimensional (EQ-5D-5L) descriptive system during the study
Body weight | 24 weeks
  Change in body weight during the study
Serum levels of 25-hydroxy-vitamin D | 24 weeks
  Change in 25-hydroxy-vitamin D during the study

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Cereda, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo; Riccardo Caccialanza, MD, Study Director — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rondanelli M, Cereda E, Klersy C, Faliva MA, Peroni G, Nichetti M, Gasparri C, Iannello G, Spadaccini D, Infantino V, Caccialanza R, Perna S. Improving rehabilitation in sarcopenia: a randomized-controlled trial utilizing a muscle-targeted food for special medical purposes. J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1535-1547. doi: 10.1002/jcsm.12532. Epub 2020 Sep 22. PMID 32961041
- [Background] Barichella M, Cereda E, Pinelli G, Iorio L, Caroli D, Masiero I, Ferri V, Cassani E, Bolliri C, Caronni S, Maggio M, Ortelli P, Ferrazzoli D, Maras A, Riboldazzi G, Frazzitta G, Pezzoli G. Muscle-targeted nutritional support for rehabilitation in patients with parkinsonian syndrome. Neurology. 2019 Jul 30;93(5):e485-e496. doi: 10.1212/WNL.0000000000007858. Epub 2019 Jul 5. PMID 31278117